CLINICAL TRIAL: NCT00001219
Title: Magnetic Resonance Imaging at 1.5 and 3.0 Tesla
Brief Title: Comparing Magnetic Resonance Imaging/Spectroscopy Techniques
Status: Terminated | Type: Observational
Why Stopped: protocol has not been used for many years and has outlived it utility
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 870091; 87-CC-0091
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Abdominal Organs - Lipodystrophy; Tumors
Keywords: MR Technology; Pulse Sequences; FDA Approved; MRI Sequences; Investigational Coils
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients undergoing MRI in the Clinical Center: All patients who, by virtue of the NIH protocol in which they are enrolled, who qualify for MRI will be eligible for participation in this protocol.

SUMMARY:
Magnetic resonance imaging (MRI) and magnetic resonance spectroscopy (MRS) are diagnostic tests that allow researchers to look at different chemical properties of tissue. Magnetic resonance imaging and spectroscopy studies can be used to gather or evaluate information about various aspects of patient s bodies or to monitor changes in the biochemistry and physiology of patient s bodies.

Unlike other diagnostic techniques (CT scan and PET scan) MRI and MRS do not use ionizing radiation. Some studies have shown that MRI is more effective at distinguishing normal parts of the anatomy from abnormal anatomy, especially in the brain. MRI has become the diagnostic test of choice for evaluating patient with multiple sclerosis.

The purpose of this study is to evaluate normal volunteers and patients with a variety of diseases with magnetic resonance imaging. Researchers will attempt different magnetic resonance imaging methods and techniques as well as different levels of magnetic strength.

DETAILED DESCRIPTION:
Background:

MRI is a constantly evolving imaging modality. Pulse sequences are often modified to improve their performance. However, many of these changes have not yet been approved by the FDA and therefore, are not considered standard of care. Some of these sequences require the use of new types of imaging coils, which are also investigational.

Objectives:

The major purpose of this protocol is to inform patients undergoing MR scans in the Clinical Center that they be scanned with MRI sequences and/or coils which may or may not be FDA approved and to get the patient s consent for this. This is not a formal research study since specific disease entities and specific pulse sequences are not studied in a systematic way. Rather, the purpose is to give NIH patients access to gradual improvements in MR technology that would otherwise not be available to them.

Eligibility:

All patients who, by virtue of the NIH protocol in which they are enrolled, qualify for MRI will be eligible for participation in this protocol.

Design:

Up to 99,999 participants will be enrolled in this study.

ELIGIBILITY:
* INCLUSION CRITERIA:
* All patients undergoing MRI in the Clinical Center.
* Patients must be able to provide informed consents.

EXCLUSION CRITERIA:

* Contraindications to MRI.
* Inability to understand consent form or consent process and the absence of a suitable guardian.
* Adults who are or may not be able to consent
* Patients in whom the scan must be performed quickly, i.e. those patients under anesthesia, anxious patients, those requiring emergency medical care, or others in which it is deemed inappropriate to prolong a study.
* Refusal to Participate.
* Pregnant women and fetuses
* Neonates

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who by virtue of the NIH protocol in which they are enrolled who qualify for MRI in the Clinical Center, are eligible to participate if (1) Stable for MRI (2) Able to understand the consent so that consent/assent can be obtained
Sampling Method: Probability Sample
Enrollment: 49946 (Actual)
Dates: Start 1987-06-18 (Actual); Primary Completion 2020-06-03 (Actual); Study Completion 2020-06-03 (Actual)

PRIMARY OUTCOMES:
Success of new sequences | 10 scan comparison
  clinically meaningful pulse sequence improvements

CONTACTS AND LOCATIONS:
Overall Officials: John A Butman, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Frank JA, Dwyer AJ, Doppman JL. Nuclear magnetic resonance imaging in oncology. Important Adv Oncol. 1987:133-74. PMID 3331379
- [Background] Roschmann P, Tischler R. Surface coil proton MR imaging at 2 T. Radiology. 1986 Oct;161(1):251-5. doi: 10.1148/radiology.161.1.3763875.
- [Background] Kim EE, Pjura G, Lowry P, Verani R, Sandler C, Flechner S, Kahan B. Cyclosporin-A nephrotoxicity and acute cellular rejection in renal transplant recipients: correlation between radionuclide and histologic findings. Radiology. 1986 May;159(2):443-6. doi: 10.1148/radiology.159.2.3515421.
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1987-CC-0091.html